CLINICAL TRIAL: NCT03735992
Title: Mind-body Medicine as a Supportive Strategy for Patients With Malignant Hematological Diseases: a Randomized Controlled Trial
Brief Title: Mind-body Medicine for Patients With Malignant Hematological Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Robert Bosch Medical Center (Other)
Responsible Party: Principal Investigator, Holger Cramer, Research Director, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBK02-17-00424
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Neoplasms
Keywords: Hematologic Neoplasms; Supportive Therapy; Fatigue; Mind-body medicine; Complementary and alternative medicine
MeSH Terms: conditions — Hematologic Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mind-body medicine group program (Experimental): Patients recieve an 11-week mind-body medicine group program including elements of mindfullness based stress reduction (MBSR), yoga, and education + treatment as usual.
  Interventions: Behavioral: Mind-body medicine group program
- Wait list (No Intervention): Treatment as usual.

INTERVENTIONS:
Behavioral: Mind-body medicine group program — The group program is mainly based on MBSR. It further integrates elements of the mind-body medicine cancer program of the Benson-Henry Mind/Body Medical Institute at Harvard Medical School which is rooted in psychoneuroendocrinology and focuses on relaxation techniques, exercise, cognitive restructuring, diet, and social support. In addition, naturopathic methods of selfregulation and self-care are incorporated.
  Arms: Mind-body medicine group program

SUMMARY:
This randomized controlled trial aims to investigate the effectiveness of a mind-body group program as a supprtivemanagement strategy for fatigue in patients with malignant hematological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant hematological diseases in complete remission after primary chemotherapy and/or radiation
* Physical and mental ability to attent 8 of 11 group units

Exclusion Criteria:

* Chemotherapy, radiation, or rehabilitation programm during the study period
* Pregnancy
* Participation in other studies with behavioral interventions during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
General Fatigue | week 12
  Multidimensional Fatigue Inventory (MFI) - General Fatigue Subscale

SECONDARY OUTCOMES:
General Fatigue | week 24
  Multidimensional Fatigue Inventory (MFI) - General Fatigue Subscale
Physical Fatigue | week 12
  Multidimensional Fatigue Inventory (MFI) - Physical Fatigue Subscale
Physical Fatigue | week 24
  Multidimensional Fatigue Inventory (MFI) - Physical Fatigue Subscale
Reduced Activity | week 12
  Multidimensional Fatigue Inventory (MFI) - Reduced Activity Subscale
Reduced Activity | week 24
  Multidimensional Fatigue Inventory (MFI) - Reduced Activity Subscale
Reduced Motivation | week 12
  Multidimensional Fatigue Inventory (MFI) - Reduced Motivation Subscale
Reduced Motivation | week 24
  Multidimensional Fatigue Inventory (MFI) - Reduced Motivation Subscale
Mental Fatigue | week 12
  Multidimensional Fatigue Inventory (MFI) - Mental Fatigue Subscale
Mental Fatigue | week 24
  Multidimensional Fatigue Inventory (MFI) - Mental Fatigue Subscale
Qaulity of life | week 12
  Functional Assessment of Cancer Therapy - General (FACT-G)
Qaulity of life | week 24
  Functional Assessment of Cancer Therapy - General (FACT-G)
Depression | week 12
  Hospital Anxiety and Depression Scale - Depression subscale (HADS-D)
Depression | week 24
  Hospital Anxiety and Depression Scale - Depression subscale (HADS-D)
Anxiety | week 12
  Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A)
Anxiety | week 24
  Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A)
Stress | week 12
  Perceived Stress Scale (PSS)
Stress | week 24
  Perceived Stress Scale (PSS)
Sleep | week 12
  Pittsburgh Sleep Quality Index (PSQI)
Sleep | week 24
  Pittsburgh Sleep Quality Index (PSQI)
Physical activity | week 12
  Motion sensor (activPAL3, Pal Technologies, Glasgow, Schottland)
Physical activity | week 24
  Motion sensor (activPAL3, Pal Technologies, Glasgow, Schottland)
Fatigability | week 12
  30-Second Chair Stand Test
Fatigability | week 24
  30-Second Chair Stand Test
Adverse Events | week 12
  Number of patients with adverse events
Adverse Events | week 24
  Number of patients with adverse events

OTHER OUTCOMES:
Treatment Expectation | week 0
  Visual Analogue Scale (VAS)
Treatment Satisfaction | week 12
  Client Satisfaction Questionnaire (CSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Director — Center for Integrative Medicine and Health, University Hospital Essen, University of Duisburg-Essen
Locations (1):
- Robert-Bosch-Krankenhaus, Abteilung für Hämatologie, Onkologie und Palliativmedizin, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request.